CLINICAL TRIAL: NCT05465187
Title: Withholding or Withdrawing of Life-sustaining Therapy in Great East French Region Intensive Care Units: a 1-month Survey
Acronym: LATA
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO22080
Record Dates: First submitted 2022-07-18; First posted 2022-07-19 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Intensive Care Units; Family's Satisfaction; Therapy Decisions
Keywords: Intensive care; family's feelings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Adults patients aged for more than 18 years old, admitted in an intensive care unit in Grand-Est region in France, for whom a decision of withholding or withdrawing of life-sustaining therapy is taken during the month of study.
  Interventions: Other: Non applicable

INTERVENTIONS:
Other: Non applicable — Non applicable

SUMMARY:
Intensive care has known an important scientists progress for the last twenty years, allowing to heal more and more severe patients. Throughout the time, population has been getting old more and more, making patients affected by several diseases.

As any medical specialty, intensive care has been confronted to these both evolutions. Thus ethical issues subsist for many years concerning rationality of cares intensity given to the patients.

Withholding or withdrawing of life-sustaining therapy represents a non-negligible part of deaths in intensive care units in France. Throughout the years, it has been more and more leading French laws, as the Clayes-Leonetti law, one of the most important and recent one, which has governed ending life patients' rights since 2016.

Thus it appears interesting to propose this study to evaluate proportion of withholding or withdrawing of life-sustaining therapy and their conditions of setting up in a maximum of intensive care units in the Grand-Est region in France in 2022 ; and to collect family's feelings concerning these decisions.

DETAILED DESCRIPTION:
Intensive care has known an important scientists progress for the last twenty years, allowing healing more and more severe patients. Throughout the time, population has been getting old more and more, making patients affected by several comorbidities.

As any medical specialty, intensive care has been confronted to these both evolutions. Thus ethical issues subsist for many years concerning rationality of cares intensity given to the patients. Depending on their age, and their comorbidities. Indeed, if cares are still possibles, disponibles and dispensables, they are not necessarily faithful.

Withholding or withdrawing of life-sustaining therapy represents a non-negligible part of deaths in intensive care units in France. In the literature, these decisions concern 8,5% to 14% of patients residents in an intensive care unit in France, with variations depending on age, so can reach 20% on patients aged more than 80 years old.

Among recent studies concerning withholding or withdrawing of life-sustaining therapy in French intensive care units, LATAREA is one of the first biggest (148 intensive care units, 7488 patients). It gives us important information about the subject. However, this study is an old one (1997), previous to Clayes-Leonetti law promulgation, which has governed ending life patients' rights since 2016. In LATAREA study, 11% of patients had measures of withholding or withdrawing of life-sustaining therapy; and mortality in intensive care units among these patients was at 78%. WLST conditions were described briefly.

A study from EPILAT group, even if more recent (2015), gives us interesting data too, but it is an ancillary study with recruitment on only 616 intensive care beds, which represented 10% of intensive care beds at the time approximately. In this study, 14% of the patients were undergoing withholding or withdrawing of life-sustaining therapy. Among notable data, we can read that an external opinion was given in less than 50% of the cases, and that less than 2% of the patients had named somebody as one's support person or had written advanced directives. It also showed that WLST percentage crossed from 8% to 30% of admissions depending on intensive care units participating.

By the way, it appears interesting to propose this study to know incidence and conditions of setting up withholding or withdrawing of life-sustaining therapy in a maximum of intensive care units in the Grand-Est region in France in 2022 ; and to collect family's feelings concerning these decisions.

ELIGIBILITY:
Inclusion criteria :

* Adults patients hospitalized in an intensive care unit in Grand-Est region in France
* For whom a decision of withholding or withdrawing of life-sustaining therapy is taken during the month of study
* Contentment of the patient or their support person collected.

Exclusion criteria :

* Patients aged less than 18 years old
* Who already have a decision of withholding or withdrawing of life-sustaining therapy taken before the beginning of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients aged for more than 18 years old hospitalized in an intensive care unit in Grand-Est region in France during the month of study, for whom a decision of withholding or withdrawing of life-sustaining therapy is taken during the month of study. Contentment of the patient or their confident person must be collected to allow inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Incidence of withholding or withdrawing of life-sustaining therapy | Day 28
  The primary outcome measure will consist in determine the part of withholding or withdrawing of life-sustaining therapy measures in Grand Est French ICU to learn about their importance. Thus we can compare it to data we know from previous studies first. Second, we can evaluate the evolution throughout the time if there is one and the impact of new laws for example.

SECONDARY OUTCOMES:
Conditions of setting up withholding or withdrawing of life-sustaining therapy | during the month of study
  Conditions can be studied by screening many data, including : data related to the intensive care unit ; data related to generalities about withholding or withdrawing of life-sustaining therapy in the center ; data related to description of population studied ; data related to the period of study ; data concerning the characteristics of the patient and measure of withholding/withdrawing of life-sustaining therapy. All data will be collected via two CRF we elaborated.
Agreement of these decisions with currently French legislation (" Claeys-Leonetti " lay, 2016) | at the inclusion of the patients in the study
  This secondary outcome measures rest on checking if the application of the measure studied in the intensive care unit is in accordance with the official law. Abuse could occur and had to be known to avoid misunderstandings and downward spiral.
Questionnaire Family Satisfaction with ICU - 24Revisited | during the month of study
  This a validated questionary to evaluate family's patient satisfaction concerning the hospitalization of their relative in the intensive care unit. More precisely, this is a global evaluation in terms of quality of cares dispensed. It is divided in two parts, included satisfaction regarding cares and satisfaction with the decision concerning patient cares in severe illness status. It ends with some demographic informations. Finally it aims is to improve fonctionnement of intensive care units.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France